CLINICAL TRIAL: NCT05256225
Title: A Phase II/III Study of Paclitaxel/Carboplatin Alone or Combined With Either Trastuzumab and Hyaluronidase-oysk (HERCEPTIN HYLECTA) or Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf (PHESGO) in HER2 Positive, Stage I-IV Endometrial Serous Carcinoma or Carcinosarcoma
Brief Title: Testing the Addition of Herceptin Hylecta or Phesgo to the Usual Chemotherapy for HER2 Positive Endometrial Serous Carcinoma or Carcinosarcoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Collaborators: NRG Oncology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-01540; NCI-2022-01540 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); NRG-GY026 (Other: NRG Oncology); NRG-GY026 (Other: CTEP); U10CA180868 (NIH)
Record Dates: First submitted 2022-02-24; First posted 2022-02-25 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-11

CONDITIONS: Endometrial Carcinoma; Endometrial Clear Cell Adenocarcinoma; Endometrial Dedifferentiated Carcinoma; Endometrial Endometrioid Adenocarcinoma; Endometrial Mixed Cell Adenocarcinoma; Endometrial Serous Adenocarcinoma; Endometrial Undifferentiated Carcinoma; Uterine Corpus Malignant Mixed Mesodermal (Mullerian) Tumor
MeSH Terms: conditions — Endometrial Neoplasms; Neoplasms | interventions — Specimen Handling; Carboplatin; Trastuzumab; pertuzumab; Paclitaxel; Taxes; Hyaluronoglucosaminidase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm I (paclitaxel, carboplatin) (Active Comparator): Patients receive paclitaxel IV over 3 hours and carboplatin IV over 30-60 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease after completion of cycle 6 may receive 4 additional cycles of this treatment at the discretion of the treating physician.
  Patients undergo ECHO or MUGA and CT throughout the study. Additionally, patients may optionally undergo blood sample collection throughout the study, vaginal brachytherapy on study, and urine sample collection prior to treatment.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Echocardiography Test; Radiation: High-Dose-Rate Vaginal Cuff Brachytherapy; Procedure: Multigated Acquisition Scan; Drug: Paclitaxel
- Arm II (paclitaxel, carboplatin, Herceptin Hylecta) (Experimental): Patients receive paclitaxel IV over 3 hours, carboplatin IV over 30-60 minutes, and trastuzumab/hyaluronidase-oysk SC over 2-5 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease after completion of cycle 6 may receive 4 additional cycles of this treatment at the discretion of the treating physician.
  MAINTENANCE: Patients receive trastuzumab/hyaluronidase-oysk SC over 2-5 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients with SD or PR may continue maintenance therapy for up to 3 years from the start of treatment.
  Patients undergo ECHO or MUGA and CT throughout the study. Additionally patients may optionally undergo blood sample collection throughout the study, vaginal brachytherapy on study, and urine sample collection prior to treatment.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Echocardiography Test; Radiation: High-Dose-Rate Vaginal Cuff Brachytherapy; Procedure: Multigated Acquisition Scan; Drug: Paclitaxel; Other: Survey Administration; Drug: Trastuzumab/Hyaluronidase-oysk
- Arm III (paclitaxel, carboplatin, Phesgo) (Experimental): See Detailed Description.
  Interventions: Procedure: Biospecimen Collection; Drug: Carboplatin; Procedure: Computed Tomography; Procedure: Echocardiography Test; Radiation: High-Dose-Rate Vaginal Cuff Brachytherapy; Drug: Hyaluronidase-zzxf/Pertuzumab/Trastuzumab; Procedure: Multigated Acquisition Scan; Drug: Paclitaxel; Other: Survey Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo blood and urine sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; JM8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Echocardiography Test — Undergo ECHO
  Other Names: EC; Echocardiography
Radiation: High-Dose-Rate Vaginal Cuff Brachytherapy — Undergo vaginal brachytherapy
  Other Names: HDR-VCB
Drug: Hyaluronidase-zzxf/Pertuzumab/Trastuzumab — Given SC
  Other Names: Pertuzumab and Trastuzumab hyaluronidase; Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; Pertuzumab/Trastuzumab/Hyaluronidase-zzxf; Phesgo
  Arms: Arm III (paclitaxel, carboplatin, Phesgo)
Procedure: Multigated Acquisition Scan — Undergo MUGA
  Other Names: Blood Pool Scan; Equilibrium Radionuclide Angiography; Gated Blood Pool Imaging; MUGA; Radionuclide Ventriculography; RNVG; SYMA Scanning; Synchronized Multigated Acquisition Scanning
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Other: Survey Administration — Ancillary studies
  Arms: Arm II (paclitaxel, carboplatin, Herceptin Hylecta); Arm III (paclitaxel, carboplatin, Phesgo)
Drug: Trastuzumab/Hyaluronidase-oysk — Given SC
  Other Names: Herceptin Hylecta; Trastuzumab and Hyaluronidase; Trastuzumab and Hyaluronidase-oysk; Trastuzumab and Recombinant Human Hyaluronidase PH20; Trastuzumab and rHuPH20; Trastuzumab-Hyaluronidase-oysk
  Arms: Arm II (paclitaxel, carboplatin, Herceptin Hylecta)

SUMMARY:
This phase III trial tests whether adding trastuzumab and hyaluronidase-oysk (Herceptin Hylecta [TM]) or pertuzumab, trastuzumab and hyaluronidase-zzxf (Phesgo [TM]) to the usual chemotherapy (paclitaxel and carboplatin) works to shrink tumors in patients with HER2 positive endometrial cancer. Trastuzumab and pertuzumab are monoclonal antibodies and forms of targeted therapy that attach to specific molecules (receptors) on the surface of tumor cells, known as HER2 receptors. When trastuzumab or pertuzumab attach to HER2 receptors, the signals that tell the cells to grow are blocked and the tumor cell may be marked for destruction by the body's immune system. Hyaluronidase is an endoglycosidase. It helps to keep pertuzumab and trastuzumab in the body longer, so that these medications will have a greater effect. Hyaluronidase also allows trastuzumab and trastuzumab/pertuzumab to be given by injection under the skin and shortens their administration time compared to trastuzumab or pertuzumab alone. Paclitaxel is a taxane and in a class of medications called antimicrotubule agents. It stops tumor cells from growing and dividing and may kill them. Carboplatin is in a class of medications known as platinum-containing compounds. It works in a way similar to the anticancer drug cisplatin, but may be better tolerated than cisplatin. Carboplatin works by killing, stopping or slowing the growth of tumor cells. Giving Herceptin Hylecta or Phesgo in combination with paclitaxel and carboplatin may shrink the tumor and prevent the cancer from coming back in patients with HER2 positive endometrial cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate the efficacy of trastuzumab and hyaluronidase-oysk (HERCEPTIN HYLECTA) and pertuzumab, trastuzumab, and hyaluronidase-zzxf (PHESGO) in combination with paclitaxel/carboplatin in patients with HER2 positive endometrial cancer.

SECONDARY OBJECTIVES:

I. To evaluate the efficacy of trastuzumab and hyaluronidase-oysk (HERCEPTIN HYLECTA) and pertuzumab, trastuzumab, and hyaluronidase-zzxf (PHESGO) in combination with paclitaxel/carboplatin in patients with HER2 positive endometrial cancer.

II. To evaluate the overall response rate (ORR) in patients with measurable disease.

III. To evaluate the duration of objective response in patients with measurable disease as assessed by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.

IV. To determine the nature, frequency and degree of toxicity as assessed by Common Terminology Criteria for Adverse Events (CTCAE) version (v.) 5.0 for each treatment arm.

V. To compare quality of life (QOL), as measured by Functional Assessment of Cancer Therapy - Endometrial Trial Outcome Index (FACT-En-TOI), in the experimental versus control arms.

VI. To compare patient-reported treatment-associated symptoms (diarrhea and rash) as measured with the Patient Reported Outcomes (PRO) - CTCAE, patient-reported fatigue as measured with the Patient Reported Outcomes Measurement Information System (PROMIS)-Fatigue short form, and worry concerning side effects of treatment as measured by the item 'bothered by side effect', in the FACT-En TOI, respectively, in the experimental and control arms.

VII. To assess the correlation of HER2 immunohistochemistry (IHC) expression and in situ hybridization (ISH) amplification with clinical outcome and response to HER2 targeted therapies.

EXPLORATORY OBJECTIVE:

I. To explore time to sustained deterioration in quality of life, as measured by a drop in the FACT-En-TOI by 6 or more points lasting for more than one PRO time point, in the experimental and control arms.

OUTLINE: Patients are randomized to 1 of 3 arms.

ARM I: Patients receive paclitaxel intravenously (IV) over 3 hours and carboplatin IV over 30-60 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with stable disease (SD) or partial response (PR) who still have measurable disease after completion of cycle 6 may receive 4 additional cycles of this treatment at the discretion of the treating physician.

ARM II: Patients receive paclitaxel IV over 3 hours, carboplatin IV over 30-60 minutes, and trastuzumab/hyaluronidase-oysk subcutaneously (SC) over 2-5 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease after completion of cycle 6 may receive 4 additional cycles of this treatment at the discretion of the treating physician.

MAINTENANCE: Patients receive trastuzumab/hyaluronidase-oysk SC over 2-5 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for up to 1 year in the absence of disease progression or unacceptable toxicity. Patients with SD or PR may continue maintenance therapy for up to 3 years from the start of treatment.

ARM III: Patients receive paclitaxel IV over 3 hours, carboplatin IV over 30-60 minutes, and pertuzumab/trastuzumab/hyaluronidase-zzxf SC over 5-8 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for 6 cycles in the absence of disease progression or unacceptable toxicity. Patients with SD or PR who still have measurable disease after completion of cycle 6 may receive 4 additional cycles of this treatment at the discretion of the treating physician.

MAINTENANCE: Patients receive pertuzumab/trastuzumab/ hyaluronidase-zzxf SC over 5 minutes on day 1 of each cycle. Cycles repeat every 3 weeks for up to 1 year in absence of disease progression or unacceptable toxicity. Patients with SD or PR may continue maintenance for up to 3 years from the start of treatment.

Patients undergo echocardiography (ECHO) or multigated acquisition scan (MUGA) and computed tomography (CT) throughout the study. Additionally, patients may optionally undergo blood sample collection throughout the study, vaginal brachytherapy on study, and urine sample collection prior to treatment.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Federation of Gynecology and Obstetrics (FIGO) 2009 stage IA-IVB, non-recurrent, chemotherapy (chemo)-naive, HER2-positive endometrial cancer. The following endometrial cancer types are eligible:

  * Serous
  * Other endometrial cancers (including clear cell, endometrioid, mixed epithelial, dedifferentiated/undifferentiated)
  * Carcinosarcoma

    * NOTE: Endometrial cancers that are mismatch repair deficient (dMMR) by IHC are not eligible
* Histologic confirmation of the original primary tumor is required. Submission of surgical pathology report (or endometrial biopsy pathology report in patients who never undergo hysterectomy) is required
* Patients must be within 8 weeks of primary surgery (or endometrial biopsy in patients who never undergo hysterectomy) at the time of study registration
* Patients may have measurable disease, non-measurable disease, or no measurable disease. In patients with measurable disease, lesions will be defined and monitored by RECIST v 1.1. Measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded). Each lesion must be >= 10 mm when measured by CT or magnetic resonance imaging (MRI). Lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* For patients with uterine-confined (stage I) disease, the tumor must be invasive into the myometrium. Any amount of myoinvasion is acceptable for eligibility. Patients with non-invasive disease, endometrial intraepithelial carcinoma alone, or disease confined to a polyp will be excluded
* All patients must have tumors that are HER2 positive as defined by American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) 2018 Breast Cancer guidelines. IHC and ISH testing will be done locally, at each participating institution and interpreted by local pathologists. In general HER2 positivity is defined as any of the following:

  * 3+ immunohistochemistry (IHC),
  * 2+ IHC with positive in situ hybridization (ISH) Alternatively, patients could be eligible if next generation sequencing (NGS) demonstrates HER2 (ERBB2) amplification. NGS testing can be performed through any designated labs as per the National Cancer Institute (NCI) MATCH/NCI Combo-MATCH trial.

Pathology report showing results of institutional HER2 testing (or NGS testing results) must be submitted.

Sites must submit all results available (IHC, ISH, and NGS)

* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2
* Age >= 18
* Platelets >= 100,000/mcl (within 14 days prior to registration)
* Absolute neutrophil count (ANC) >= 1,500/mcl (within 14 days prior to registration)
* Creatinine =< 1.5 x institutional/laboratory upper limit of normal (ULN) or estimated Glomerular filtration rate (eGFR) >= 50 mL/min using either the Cockcroft-Gault equation, the Modification of Diet in Renal Disease Study, or as reported in the comprehensive metabolic panel/basic metabolic panel (eGFR) (within 14 days prior to registration)
* Total serum bilirubin level =< 1.5 x ULN (patients with known Gilbert's disease who have bilirubin level =< 3 x ULN may be enrolled) (within 14 days prior to registration)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 3 x ULN (within 14 days prior to registration)
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of registration are eligible for this trial
* Although the uterus will have been removed in the vast majority of patients, for patients of child-bearing potential: negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required. Patients will be considered of non-reproductive potential if they are either:

  * Postmenopausal (defined as at least 12 months with no menses without an alternative medical cause; in women < 45 years of age, a high follicle stimulating hormone [FSH] level in the postmenopausal range may be used to confirm a postmenopausal state in women not using hormonal contraception or hormonal replacement therapy. In the absence of 12 months of amenorrhea, a single FSH measurement is insufficient); OR
  * Have had a hysterectomy and/or bilateral oophorectomy, bilateral salpingectomy or bilateral tubal ligation/occlusion at least 6 weeks prior to registration
  * Have a congenital or acquired condition that prevents childbearing
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with evidence of chronic hepatitis B virus (HBV) infection must have an undetectable HBV viral load on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* The patient or a legally authorized representative must provide study-specific informed consent prior to study entry and, for patients treated in the United States (U.S.), authorization permitting release of personal health information

Exclusion Criteria:

* Prior Therapy:

  * Patients must NOT have received prior chemotherapy, biologic therapy, or targeted therapy for treatment of endometrial carcinoma
  * Patients must NOT have received prior radiation therapy for treatment of endometrial carcinoma. Prior radiation includes external beam pelvic radiation therapy, external beam extended field pelvic/para-aortic radiation therapy, and/or intravaginal brachytherapy

    * NOTE: Vaginal brachytherapy for treatment of endometrial cancer is permitted during study treatment. Planned use of vaginal brachytherapy must be declared at time of registration
  * Patients may have received prior hormonal therapy for treatment of endometrial carcinoma. All hormonal therapy must be discontinued at least one week prior to registration
* Patients may not have a planned interval cytoreduction or hysterectomy, prior to documentation of progression, after study registration
* Patients may not have planned external beam radiotherapy, prior to documentation of progression, after study registration
* Significant cardiovascular disease including:

  * Uncontrolled hypertension, defined as systolic > 150 mm Hg or diastolic > 90 mm Hg despite antihypertensive medications
  * Myocardial infarction or unstable angina within 6 months prior to registration
  * New York Heart Association functional classification II, III or IV
  * Serious cardiac arrhythmia requiring medication. This does not include asymptomatic, atrial fibrillation with controlled ventricular rate
* Significant lung disease: dyspnea at rest grade 2 or greater (resulting from extensive tumor involvement or other causes), pneumonitis grade 2 or greater, interstitial lung disease grade 2 or greater, idiopathic pulmonary fibrosis, cystic fibrosis, Aspergillosis, active tuberculosis, or history of opportunistic infections (pneumocystis pneumonia or cytomegalovirus pneumonia)
* Patients with uncontrolled intercurrent illness including, but not limited to: ongoing or active infection (except for uncomplicated urinary tract infection), uncontrolled interstitial lung disease, symptomatic congestive heart failure, or psychiatric illness/social situations that would limit compliance with study requirements
* Treatment with strong CYP2C8 or CYP3A4 inhibitors or inducers within 14 days or 5 drug-elimination half-lives, whichever is longer, prior to registration
* Women who are unwilling to discontinue nursing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-11-16 (Actual); Primary Completion 2027-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | From study entry to time of progression or death, whichever occurs first, or date of last contact if neither progression nor death has occurred, assessed up to 5 years from randomization
  At the end of Phase 2 analysis, if both experimental arms demonstrate superiority to the reference, the experimental arms will be compared to each other.
Overall survival | From study entry to time of death or the date of last contact, assessed up to 5 years from randomization
  If both experimental arms demonstrate superiority to the reference arm, the experimental arms will be compared to each other.
Incidence of dose limiting toxicities | Up to end of cycle 3 (week 12)
  A dose limiting toxicity is any treatment-related adverse event requiring permanent discontinuation of the experimental therapy prior to the completion of treatment cycle 3.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Within 12 months of initiating maintenance therapy
  Defined as the binomial proportion of evaluable patients with a best overall response of complete response or partial response (by Response Evaluation Criteria in Solid Tumors 1.1) within 12 months of initiating maintenance therapy. Responses reported by the treating physician will be used for these analyses. The ORR estimates by treatment arm will be supported by their 2-sided, 95% Wilson-Score confidence intervals (Wilson, 1927; Agresti, 1998). The relative odds of response in each experimental group (versus [vs] the reference group) will be estimated using a multivariable logistic regression model specified with main effects for the treatment groups and covariate adjustments for the stratification factors reported at baseline.
Duration of objective response | From documentation of either PR or CR until disease progression or death, whichever is observed first, assessed up to 5 years from randomization
  Treatment group differences in response duration will be graphed using Kaplan-Meier methods and compared using logrank tests, stratified by the minimization factors defined at randomization. The relative hazards of progression or death in each experimental group (vs the reference group) will be estimated using a multivariable proportional hazards regression model specified with main effects for the treatment indicators and covariate adjustments for the stratification factors reported at baseline.
Incidence of adverse events (AEs) | Up to 5 years from randomization
  The nature, frequency, and degree of toxicity will be tabulated at the System Organ Class and AE-specific term levels using Common Terminology Criteria version 5.0. Each patient will be represented according to the maximum grade observed for each term. Tabulations will show the number and percentage of patients by maximum grade, within the treatment group received, regardless of the randomized treatment assignment.
HER2 expression | Up to 5 years from randomization
  Correlation of HER2 immunohistochemistry expression and in situ hybridization amplification with clinical outcome and response to HER2 targeted therapies will be explored.
Quality of life (QoL) | Up to 5 years from randomization
  Measured by Functional Assessment of Cancer Therapy - Endometrial Trial Outcome Index.

OTHER OUTCOMES:
QoL deterioration | Baseline up to 5 years
  The deterioration in QoL will be measured by a drop of >= 6 points in the FACT-En TOI score from baseline and lasting for more than one patient reported outcome time point in experimental and control arms.

CONTACTS AND LOCATIONS:
Overall Officials: Britt K Erickson, Principal Investigator — NRG Oncology
Locations (407):
- United States (403):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - Alaska Women's Cancer Care, Anchorage, Alaska
  - Banner University Medical Center - Tucson, Tucson, Arizona
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Sutter Auburn Faith Hospital, Auburn, California
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - John Muir Medical Center-Concord, Concord, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - City of Hope Seacliff, Huntington Beach, California
  - UCI Health - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Kaiser Permanente-Irvine, Irvine, California
  - City of Hope at Long Beach Elm, Long Beach, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Memorial Medical Center, Modesto, California
  - Palo Alto Medical Foundation-Gynecologic Oncology, Mountain View, California
  - Saint Joseph Hospital - Orange, Orange, California
  - UC Irvine Health/Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Kaiser Permanente - Panorama City, Panorama City, California
  - Kaiser Permanente-Riverside, Riverside, California
  - Sutter Roseville Medical Center, Roseville, California
  - Sutter Medical Center Sacramento, Sacramento, California
  - University of California Davis Comprehensive Cancer Center, Sacramento, California
  - California Pacific Medical Center-Pacific Campus, San Francisco, California
  - Palo Alto Medical Foundation-Santa Cruz, Santa Cruz, California
  - Palo Alto Medical Foundation-Sunnyvale, Sunnyvale, California
  - City of Hope Upland, Upland, California
  - John Muir Medical Center-Walnut Creek, Walnut Creek, California
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UCHealth - Cherry Creek, Denver, Colorado
  - AdventHealth Porter, Denver, Colorado
  - Grand Valley Oncology, Grand Junction, Colorado
  - Banner North Colorado Medical Center, Greeley, Colorado
  - UCHealth Highlands Ranch Hospital, Highlands Ranch, Colorado
  - Banner North Colorado Medical Center - Loveland Campus, Loveland, Colorado
  - Danbury Hospital, Danbury, Connecticut
  - Smilow Cancer Hospital-Derby Care Center, Derby, Connecticut
  - Smilow Cancer Hospital Care Center-Fairfield, Fairfield, Connecticut
  - Smilow Cancer Hospital Care Center at Glastonbury, Glastonbury, Connecticut
  - Smilow Cancer Hospital Care Center at Greenwich, Greenwich, Connecticut
  - Smilow Cancer Hospital Care Center - Guilford, Guilford, Connecticut
  - Smilow Cancer Hospital Care Center at Saint Francis, Hartford, Connecticut
  - Yale University, New Haven, Connecticut
  - Yale-New Haven Hospital North Haven Medical Center, North Haven, Connecticut
  - Norwalk Hospital, Norwalk, Connecticut
  - Smilow Cancer Hospital Care Center at Long Ridge, Stamford, Connecticut
  - Smilow Cancer Hospital-Torrington Care Center, Torrington, Connecticut
  - Smilow Cancer Hospital Care Center-Trumbull, Trumbull, Connecticut
  - Smilow Cancer Hospital-Waterbury Care Center, Waterbury, Connecticut
  - Smilow Cancer Hospital Care Center - Waterford, Waterford, Connecticut
  - Helen F Graham Cancer Center, Newark, Delaware
  - Medical Oncology Hematology Consultants PA, Newark, Delaware
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - George Washington University Medical Center, Washington D.C., District of Columbia
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - Sarasota Memorial Hospital-Venice, N. Venice, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Florida Cancer Specialists - Sarasota Downtown, Sarasota, Florida
  - First Physicians Group-Sarasota, Sarasota, Florida
  - Sarasota Memorial Hospital, Sarasota, Florida
  - Florida Cancer Specialists - Venice Pinebrook, Venice, Florida
  - Grady Health System, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia
  - Augusta University Medical Center, Augusta, Georgia
  - Emory Decatur Hospital, Decatur, Georgia
  - Lewis Cancer and Research Pavilion at Saint Joseph's/Candler, Savannah, Georgia
  - Queen's Medical Center, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Saint Alphonsus Cancer Care Center-Boise, Boise, Idaho
  - Saint Luke's Cancer Institute - Boise, Boise, Idaho
  - Saint Alphonsus Cancer Care Center-Caldwell, Caldwell, Idaho
  - Kootenai Health - Coeur d'Alene, Coeur d'Alene, Idaho
  - Saint Luke's Cancer Institute - Fruitland, Fruitland, Idaho
  - Saint Luke's Cancer Institute - Meridian, Meridian, Idaho
  - Saint Alphonsus Cancer Care Center-Nampa, Nampa, Idaho
  - Saint Luke's Cancer Institute - Nampa, Nampa, Idaho
  - Kootenai Clinic Cancer Services - Post Falls, Post Falls, Idaho
  - Kootenai Clinic Cancer Services - Sandpoint, Sandpoint, Idaho
  - Saint Luke's Cancer Institute - Twin Falls, Twin Falls, Idaho
  - Northwest Community Hospital, Arlington Heights, Illinois
  - Rush-Copley Medical Center, Aurora, Illinois
  - Centralia Oncology Clinic, Centralia, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Rush MD Anderson Cancer Center, Chicago, Illinois
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Carle at The Riverfront, Danville, Illinois
  - Cancer Care Specialists of Illinois - Decatur, Decatur, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Northwestern Medicine Cancer Center Kishwaukee, DeKalb, Illinois
  - Carle Physician Group-Effingham, Effingham, Illinois
  - Crossroads Cancer Center, Effingham, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Northwestern Medicine Cancer Center Delnor, Geneva, Illinois
  - NorthShore University HealthSystem-Glenbrook Hospital, Glenview, Illinois
  - Northwestern Medicine Glenview Outpatient Center, Glenview, Illinois
  - Northwestern Medicine Grayslake Outpatient Center, Grayslake, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - NorthShore University HealthSystem-Highland Park Hospital, Highland Park, Illinois
  - Sudarshan K Sharma MD Limited-Gynecologic Oncology, Hinsdale, Illinois
  - Northwestern Medicine Lake Forest Hospital, Lake Forest, Illinois
  - Carle Physician Group-Mattoon/Charleston, Mattoon, Illinois
  - UC Comprehensive Cancer Center at Silver Cross, New Lenox, Illinois
  - Carle Cancer Institute Normal, Normal, Illinois
  - Cancer Care Center of O'Fallon, O'Fallon, Illinois
  - Northwestern Medicine Orland Park, Orland Park, Illinois
  - University of Chicago Medicine-Orland Park, Orland Park, Illinois
  - UW Health Carbone Cancer Center Rockford, Rockford, Illinois
  - Southern Illinois University School of Medicine, Springfield, Illinois
  - Springfield Clinic, Springfield, Illinois
  - Springfield Memorial Hospital, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Northwestern Medicine Cancer Center Warrenville, Warrenville, Illinois
  - Rush-Copley Healthcare Center, Yorkville, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Northwest Cancer Center - Main Campus, Crown Point, Indiana
  - UChicago Medicine Northwest Indiana, Crown Point, Indiana
  - Northwest Oncology LLC, Dyer, Indiana
  - Goshen Center for Cancer Care, Goshen, Indiana
  - Northwest Cancer Center - Hobart, Hobart, Indiana
  - Saint Mary Medical Center, Hobart, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - Franciscan Health Indianapolis, Indianapolis, Indiana
  - Ascension Saint Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Saint Catherine Hospital, Indianapolis, Indiana
  - Franciscan Saint Elizabeth Health - Lafayette East, Lafayette, Indiana
  - Franciscan Health Mooresville, Mooresville, Indiana
  - The Community Hospital, Munster, Indiana
  - Women's Diagnostic Center - Munster, Munster, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northwest Cancer Center - Valparaiso, Valparaiso, Indiana
  - Mary Greeley Medical Center, Ames, Iowa
  - McFarland Clinic - Ames, Ames, Iowa
  - McFarland Clinic - Boone, Boone, Iowa
  - Heartland Oncology and Hematology LLP, Council Bluffs, Iowa
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MEJ, Council Bluffs, Iowa
  - McFarland Clinic - Trinity Cancer Center, Fort Dodge, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - McFarland Clinic - Jefferson, Jefferson, Iowa
  - McFarland Clinic - Marshalltown, Marshalltown, Iowa
  - Saint Elizabeth Healthcare Edgewood, Edgewood, Kentucky
  - Baptist Health Lexington, Lexington, Kentucky
  - Baptist Health Louisville, Louisville, Kentucky
  - LSU Health Baton Rouge-North Clinic, Baton Rouge, Louisiana
  - Our Lady of the Lake Physician Group, Baton Rouge, Louisiana
  - Our Lady of the Lake Medical Oncology, Baton Rouge, Louisiana
  - Ochsner Hematology Oncology North Shore - Covington (West Region), Covington, Louisiana
  - West Jefferson Medical Center, Marrero, Louisiana
  - East Jefferson General Hospital, Metairie, Louisiana
  - LSU Healthcare Network / Metairie Multi-Specialty Clinic, Metairie, Louisiana
  - University Medical Center New Orleans, New Orleans, Louisiana
  - Ochsner Baptist Medical Center, New Orleans, Louisiana
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - Harold Alfond Center for Cancer Care, Augusta, Maine
  - MaineHealth Maine Medical Center- Scarborough, Scarborough, Maine
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Sinai Hospital of Baltimore, Baltimore, Maryland
  - MedStar Franklin Square Medical Center/Weinberg Cancer Institute, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - William E Kahlert Regional Cancer Center/Sinai Hospital, Westminster, Maryland
  - Baystate Medical Center, Springfield, Massachusetts
  - University of Michigan Rogel Cancer Center, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Brighton, Brighton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Canton, Canton, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology - Chelsea Hospital, Chelsea, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Weisberg Cancer Treatment Center, Farmington Hills, Michigan
  - Corewell Health Farmington Hills Hospital, Farmington Hills, Michigan
  - Cancer Hematology Centers - Flint, Flint, Michigan
  - Genesee Hematology Oncology PC, Flint, Michigan
  - Genesys Hurley Cancer Institute, Flint, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Trinity Health Grand Rapids Hospital, Grand Rapids, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Beacon Kalamazoo Cancer Center, Kalamazoo, Michigan
  - Trinity Health Saint Mary Mercy Livonia Hospital, Livonia, Michigan
  - Trinity Health Muskegon Hospital, Muskegon, Michigan
  - Corewell Health Lakeland Hospitals - Niles Hospital, Niles, Michigan
  - Cancer and Hematology Centers of Western Michigan - Norton Shores, Norton Shores, Michigan
  - Trinity Health Saint Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Corewell Health Reed City Hospital, Reed City, Michigan
  - Corewell Health William Beaumont University Hospital, Royal Oak, Michigan
  - MyMichigan Medical Center Saginaw, Saginaw, Michigan
  - Oncology Hematology Associates of Saginaw Valley PC, Saginaw, Michigan
  - Corewell Health Lakeland Hospitals - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - Corewell Health Lakeland Hospitals - Saint Joseph Hospital, Saint Joseph, Michigan
  - MyMichigan Medical Center Tawas, Tawas City, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Corewell Health Beaumont Troy Hospital, Troy, Michigan
  - Saint Mary's Oncology/Hematology Associates of West Branch, West Branch, Michigan
  - University of Michigan Health - West, Wyoming, Michigan
  - Trinity Health IHA Medical Group Hematology Oncology Ann Arbor Campus, Ypsilanti, Michigan
  - Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Avera Cancer Institute at Marshall, Marshall, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - University of Minnesota/Masonic Cancer Center, Minneapolis, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Minnesota Oncology Hematology PA-Woodbury, Woodbury, Minnesota
  - MU Health - University Hospital/Ellis Fischel Cancer Center, Columbia, Missouri
  - Phelps Health Delbert Day Cancer Institute, Rolla, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Mercy Hospital South, St Louis, Missouri
  - Mercy Hospital Saint Louis, St Louis, Missouri
  - Community Hospital of Anaconda, Anaconda, Montana
  - Billings Clinic Cancer Center, Billings, Montana
  - Saint Vincent Frontier Cancer Center, Billings, Montana
  - Intermountain Health West End Clinic, Billings, Montana
  - Bozeman Health Deaconess Hospital, Bozeman, Montana
  - Benefis Sletten Cancer Institute, Great Falls, Montana
  - Logan Health Medical Center, Kalispell, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Community Medical Center, Missoula, Montana
  - Nebraska Cancer Specialists/Oncology Hematology West PC - MECC, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - OptumCare Cancer Care at Seven Hills, Henderson, Nevada
  - OptumCare Cancer Care at Charleston, Las Vegas, Nevada
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - OptumCare Cancer Care at Fort Apache, Las Vegas, Nevada
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Monmouth Medical Center Southern Campus, Lakewood, New Jersey
  - Saint Barnabas Medical Center, Livingston, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Virtua Samson Cancer Center, Moorestown, New Jersey
  - Jersey Shore Medical Center, Neptune City, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Riverview Medical Center/Booker Cancer Center, Red Bank, New Jersey
  - Sidney Kimmel Cancer Center Washington Township, Sewell, New Jersey
  - Robert Wood Johnson University Hospital Somerset, Somerville, New Jersey
  - Community Medical Center, Toms River, New Jersey
  - Virtua Voorhees, Voorhees Township, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - Presbyterian Rust Medical Center/Jorgensen Cancer Center, Rio Rancho, New Mexico
  - Women's Cancer Care Associates LLC, Albany, New York
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - NYU Langone Hospital - Long Island, Mineola, New York
  - Mount Sinai Chelsea, New York, New York
  - Laura and Isaac Perlmutter Cancer Center at NYU Langone, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Wilmot Cancer Institute at Webster, Webster, New York
  - Duke Cancer Center Cary, Cary, North Carolina
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - ECU Health Medical Center, Greenville, North Carolina
  - Hayworth Cancer Center, High Point, North Carolina
  - Duke Women's Cancer Care Raleigh, Raleigh, North Carolina
  - Novant Health New Hanover Regional Medical Center, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Broadway Medical Center, Fargo, North Dakota
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - UHHS-Chagrin Highlands Medical Center, Beachwood, Ohio
  - Strecker Cancer Center-Belpre, Belpre, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Miami Valley Hospital South, Centerville, Ohio
  - Geauga Hospital, Chardon, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - Good Samaritan Hospital - Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - Mount Carmel East Hospital, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - The Mark H Zangmeister Center, Columbus, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Miami Valley Hospital North, Dayton, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Miami Valley Cancer Care and Infusion, Greenville, Ohio
  - Mount Carmel Grove City Hospital, Grove City, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Saint Rita's Medical Center, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Memorial Hospital, Marysville, Ohio
  - UH Seidman Cancer Center at Lake Health Mentor Campus, Mentor, Ohio
  - Knox Community Hospital, Mount Vernon, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Mercy Health - Perrysburg Hospital, Perrysburg, Ohio
  - Southern Ohio Medical Center, Portsmouth, Ohio
  - Springfield Regional Cancer Center, Springfield, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - Mercy Health - Saint Vincent Hospital, Toledo, Ohio
  - Mercy Health - Saint Anne Hospital, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - UH Seidman Cancer Center at Saint John Medical Center, Westlake, Ohio
  - Genesis Healthcare System Cancer Care Center, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Mercy Hospital Oklahoma City, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Providence Cancer Institute Clackamas Clinic, Clackamas, Oregon
  - Providence Newberg Medical Center, Newberg, Oregon
  - Saint Alphonsus Cancer Care Center-Ontario, Ontario, Oregon
  - Legacy Good Samaritan Hospital and Medical Center, Portland, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Oregon Health and Science University, Portland, Oregon
  - Legacy Meridian Park Hospital, Tualatin, Oregon
  - Lehigh Valley Hospital-Cedar Crest, Allentown, Pennsylvania
  - Saint Luke's Cancer Center - Allentown, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Pocono Medical Center, East Stroudsburg, Pennsylvania
  - Saint Luke's Hospital-Anderson Campus, Easton, Pennsylvania
  - Saint Vincent Hospital, Erie, Pennsylvania
  - Lehigh Valley Hospital-Hazleton, Hazleton, Pennsylvania
  - Jefferson Hospital, Jefferson Hills, Pennsylvania
  - Riddle Memorial Hospital, Media, Pennsylvania
  - Forbes Hospital, Monroeville, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Saint Luke's Hospital - Upper Bucks Campus, Quakertown, Pennsylvania
  - Chester County Hospital, West Chester, Pennsylvania
  - Wexford Health and Wellness Pavilion, Wexford, Pennsylvania
  - Asplundh Cancer Pavilion, Willow Grove, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Smilow Cancer Hospital Care Center - Westerly, Westerly, Rhode Island
  - Saint Joseph's/Candler - Bluffton Campus, Bluffton, South Carolina
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute-Aberdeen, Aberdeen, South Dakota
  - Rapid City Regional Hospital, Rapid City, South Dakota
  - Sanford Cancer Center Oncology Clinic, Sioux Falls, South Dakota
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - The West Clinic - Wolf River, Germantown, Tennessee
  - Dell Seton Medical Center at The University of Texas, Austin, Texas
  - University of Texas at Austin, Austin, Texas
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas
  - Tarrant County Hospital District/JPS Health Network, Fort Worth, Texas
  - UT Southwestern/Simmons Cancer Center-Fort Worth, Fort Worth, Texas
  - Houston Methodist Hospital, Houston, Texas
  - Memorial Hermann Texas Medical Center, Houston, Texas
  - Methodist Willowbrook Hospital, Houston, Texas
  - Houston Methodist West Hospital, Houston, Texas
  - Houston Methodist Saint John Hospital, Nassau Bay, Texas
  - UT Southwestern Clinical Center at Richardson/Plano, Richardson, Texas
  - Houston Methodist Sugar Land Hospital, Sugar Land, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - South Jordan Health Center, South Jordan, Utah
  - University of Virginia Cancer Center, Charlottesville, Virginia
  - Henrico Doctor's Hospital, Richmond, Virginia
  - VCU Massey Cancer Center at Stony Point, Richmond, Virginia
  - VCU Massey Comprehensive Cancer Center, Richmond, Virginia
  - Carilion Roanoke Memorial Hospital, Roanoke, Virginia
  - Swedish Cancer Institute-Edmonds, Edmonds, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - Legacy Salmon Creek Hospital, Vancouver, Washington
  - West Virginia University Charleston Division, Charleston, West Virginia
  - West Virginia University Healthcare, Morgantown, West Virginia
  - Marshfield Medical Center-EC Cancer Center, Eau Claire, Wisconsin
  - Saint Vincent Hospital Cancer Center Green Bay, Green Bay, Wisconsin
  - Saint Vincent Hospital Cancer Center at Saint Mary's, Green Bay, Wisconsin
  - Gundersen Lutheran Medical Center, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center - Eastpark Medical Center, Madison, Wisconsin
  - University of Wisconsin Carbone Cancer Center - University Hospital, Madison, Wisconsin
  - Marshfield Medical Center-Marshfield, Marshfield, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin
  - Marshfield Medical Center - Minocqua, Minocqua, Wisconsin
  - ProHealth D N Greenwald Center, Mukwonago, Wisconsin
  - Cancer Center of Western Wisconsin, New Richmond, Wisconsin
  - ProHealth Oconomowoc Memorial Hospital, Oconomowoc, Wisconsin
  - Saint Vincent Hospital Cancer Center at Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Medical Center-Rice Lake, Rice Lake, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sheboygan, Sheboygan, Wisconsin
  - Sheboygan Physicians Group, Sheboygan, Wisconsin
  - Marshfield Medical Center-River Region at Stevens Point, Stevens Point, Wisconsin
  - Saint Vincent Hospital Cancer Center at Sturgeon Bay, Sturgeon Bay, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
  - Marshfield Medical Center - Weston, Weston, Wisconsin
- Centro Comprensivo de Cancer de UPR, San Juan, Puerto Rico
- South Korea (3):
  - Keimyung University-Dongsan Medical Center, Dalseo-gu, Daegu
  - Samsung Changwon Hospital, Seoul, Gyeongsangnam-do
  - Gangnam Severance Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page
URL: https://grants.nih.gov/policy/sharing.htm

REFERENCES:
- [Derived] Secord AA, Powell MA, McAlpine J. Molecular Characterization and Clinical Implications of Endometrial Cancer. Obstet Gynecol. 2025 Nov 1;146(5):660-671. doi: 10.1097/AOG.0000000000006080. Epub 2025 Sep 18. PMID 40966692